CLINICAL TRIAL: NCT06105086
Title: Risk Analysis Interview IVDR 2023
Acronym: RAI-IVDR23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Johan Guns, Prof., Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23353_RAI-IVDR23
Record Dates: First submitted 2023-10-10; First posted 2023-10-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Risk Variables
Keywords: IH-IVD; in-house tests; IVDR 2017/746; Semi-structured interview; Risk analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- medical doctors and clinical laboratory managers (Experimental): Semi-structured interviews
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Participants will be asked pre-defined questions and are allowed to elaborate on the subject.

SUMMARY:
The objective of this research project is to design a risk-based model to decide when clinical performance studies should be performed on in-house developed in vitro diagnostic tests (IH-IVDs) in compliance with the European in vitro diagnostics regulation (EU IVDR 2017/746). To construct the dataset, semi-structured interviews will be conducted to assess the clinical hazards of the in-house in vitro diagnostic test assessments, their degree of significance and their importance with respect to clinical performance, as determined by the opinions of field specialists.

DETAILED DESCRIPTION:
The project's intervention involves conducting semi-structured interviews with clinical laboratory managers and medical professionals. The estimated number of participants for this study is 30. Various In-house in vitro diagnostic tests (IH-IVDs) will be selected, that are classified under different categories according to the risk management in the new IVDR. Two interviews will be conducted for each test. These interviews will engage a laboratory technician and a medical expert specialized in that particular test. The purpose of these interviews is to gather data on the variables that contribute to the risks of IH-IVDs and their impact on clinical diagnosis and patient outcomes. The obtained results will be applied in creating a decision tree using a pre-validated algorithm. The semi-structured interviews feature pre-determined questions that allow participants to share their experiences and opinions within their area of expertise. Each interview is expected to last between thirty minutes to an hour. If consent is given, the interviews will be recorded but not published or shared. In accordance with the confidentiality policy, all data collected will be kept anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Work relation with the medical field/hospital
* Achieved a master degree or higher
* Compatible to take an interview independently

Exclusion Criteria:

/

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Risk attributes of the in-house in vitro diagnostic tests measured with semi-structured interviews | 1 hour
  Risk attributes of the in-house in vitro diagnostic tests are the variables that have an impact on the clinical diagnosis and patient outcome. This will be measured with a semi-structured interview with medical doctors and laboratory managers.
risk impact of the in-house in vitro diagnostic tests measured with semi-structured interviews | 1 hour
  With the opinions and experience of professionals in the field of interest, the risk impact of the in-house in vitro diagnostic tests will be measured with semi-structured interviews. The impact defines the severity or importance of the risk attributes.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Guns, Prof., Principal Investigator — UZ Brussel Laboratorium Kwaliteit
Locations (1):
- UZ brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Everything that potentially is going to be shared is anonymous.